CLINICAL TRIAL: NCT02934412
Title: A Phase I, Randomized, Double-blind, Placebo-controlled, Single Dose Escalation Study to Investigate Safety and Pharmacokinetics of SHR-1314 in Healthy Subjects
Brief Title: A Study of SHR-1314 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atridia Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: SHR-1314-A101
Record Dates: First submitted 2016-09-20; First posted 2016-10-17 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- SHR-1314 20mg (Experimental): 20mg SHR-1314 or placebo is administered subcutaneously to healthy subjects
  Interventions: Drug: SHR-1314; Drug: placebo
- SHR-1314 40mg (Experimental): 40mg SHR-1314 or placebo is administered subcutaneously to healthy subjects
  Interventions: Drug: SHR-1314; Drug: placebo
- SHR-1314 80mg (Experimental): 80mg SHR-1314 or placebo is administered subcutaneously to healthy subjects
  Interventions: Drug: SHR-1314; Drug: placebo
- SHR-1314 160mg (Experimental): 160mg SHR-1314 or placebo is administered subcutaneously to healthy subjects
  Interventions: Drug: SHR-1314; Drug: placebo
- SHR-1314 240mg (Experimental): 240mg SHR-1314 or placebo is administered subcutaneously to healthy subjects
  Interventions: Drug: SHR-1314; Drug: placebo

INTERVENTIONS:
Drug: SHR-1314 — Single subcutaneous injection of SHR-1314 at 5 dose levels (20mg, 40mg, 80mg, 160mg, and 240mg) in healthy subjects.
Drug: placebo — Single subcutaneous injection of placebo at 5 dose levels (20mg, 40mg, 80mg, 160mg, and 240mg) in healthy subjects.

SUMMARY:
This is a randomized, double-blind, placebo-controlled, single dose escalating, study in 5 sequential cohorts to investigate the effect of a single s.c. injection of SHR-1314 at 5 dose levels (20mg, 40mg, 80mg, 160mg, and 240mg) in healthy subjects. Each cohort will consist of 6 subjects receiving active drug and 2 subjects receiving placebo, for a total of approximately 40 subjects dosed at one study site.

DETAILED DESCRIPTION:
This study will consist of a 27-day screening period (Days -28 to -2), clinic check-in (Day -1), a treatment day (Day 1), a 10-week treatment period and a study completion evaluation (Day 71) as shown in above figure.

A review of blinded interim PK data will be conducted by the Safety Review Committee (SRC) to confirm the study sampling schedule captures the full PK profile of SHR-1314. This interim analysis will be conducted for Cohort 1 and may be conducted for subsequent cohorts if serum SHR-1314 concentrations in Cohort 1 or any of the subsequent cohorts are below the limit of quantification of the assay preventing evaluation of the PK profile.

The expected duration of participation for each subject will be up to 99 days. Subjects who are withdrawn for reasons other than safety may be replaced at the discretion of the sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent before any study assessment is performed.
2. Male or female between the ages of 18 and 55 years (inclusive) at screening,
3. Good general health as defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination including measurement of vital signs, 12-lead ECG, and clinical laboratory tests. (Evaluations must be considered "not clinically significant (NCS)" if outside of the reference range).
4. Body Mass Index (BMI) of 18 to 30 kg/m2 (inclusive), and a total body weight ≥50 kg at screening.
5. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures as specified in the protocol.

Exclusion Criteria:

1. Subjects who are investigational site staff members or subjects who are Sponsor employees directly involved in the conduct of the study.
2. Use of other investigational drugs within 5 half-lives of screening, or within 30 days of screening (for small molecules), or until the expected pharmacodynamic effect has returned to baseline (for biologics), whichever is longer.
3. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin laboratory test at screening or Day -1.
4. Females of child-bearing potential (defined as all females physiologically capable of becoming pregnant) and males who are unwilling or unable to use effective contraception during the study and until 2 months after drug administration (approximately 5 half-lives). Effective contraception is defined use of two of the following methods of contraception:

   * Barrier method: Condom or Occlusive cap (diaphragm or cervical/vault caps).
   * Female sterilization: have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
   * Male sterilization
   * Use of established oral, injected or implanted hormonal methods of contraception,
   * Use of an intrauterine device or intrauterine system.
5. Blood donation of approximately 500 mL within 56 days prior to dosing on Day 1 and for the duration of the study.
6. A positive urine drug screen at screening and Day -1.
7. History of regular alcohol consumption exceeding 14 drinks/week for females or 21 drinks/week for males (1 drink = 100 mL of wine or 360 mL of beer or 45 mL of hard liquor) within 6 months of screening.
8. Use of tobacco or nicotine containing products (including e-cigarettes) at any time within six months before screening and for the duration of the study.
9. History of hypersensitivity to any of the study biologics, drugs or to drugs of similar chemical classes.
10. History of malignancy of any organ system, treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
11. History or complication of tuberculosis.
12. Has a clinically significant abnormality on the screening chest x-ray that, in the opinion of the investigator, could affect the subject's safety or ability to participate in the study; including, but not limited to, evidence of previous exposure to tuberculosis.
13. History of immunodeficiency diseases, including a positive human immunodeficiency virus (HIV) test result at screening.
14. Positive hepatitis B or hepatitis C test result at Screening
15. Recent (within the last 3 years) and/or recurrent history of acute or chronic bronchospastic pulmonary disease (including asthma and chronic obstructive pulmonary disease, treated or not treated).
16. Use of live vaccines (attenuated) within 3 months before study Day 1 or at any time during the study.
17. Evidence of latent tuberculosis by QuantiFERON screening.
18. Use of any of the following, unless agreed as non-clinically relevant by the Investigator and the Sponsor:

    1. Prescription medication within four weeks prior to dosing on Day 1
    2. Over-the-counter medication (excluding paracetamol) within seven days prior to the treatment day. Paracetamol use must be limited to 2 g per day and no more than three days usage in the four weeks prior to dosing on Day 1
    3. Vitamin therapy or dietary supplements within seven days prior to dosing on Day 1 and for the duration of the study
    4. Herbal supplements within 28 days prior to the dosing on Day 1 and for the duration of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-08-22 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | 70 days

SECONDARY OUTCOMES:
Serum concentrations of SHR01314 | 70 days
Serum anti-drug antibodies | 70 days

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Farinola, B.Sc,BMBS, Principal Investigator — Royal Adelaide Hospital
Locations (1):
- Atridia Pty Limited, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No